CLINICAL TRIAL: NCT05424731
Title: Viaskin® Peanut (DBV712) Compassionate Use in Peanut-allergic Children Previously Enrolled in a DBV712 Clinical Study
Brief Title: Expanded Access Protocol of Viaskin® Peanut (DBV712) in Peanut-allergic Children
Status: Available | Type: Expanded Access
Sponsor: DBV Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: V712-EAP02
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Peanut Allergy
Keywords: EPIT; Epicutaneous; Immunotherapy; Viaskin
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Combination Product: DBV712 250 mcg — Daily epicutaneous delivery.
  Other Names: Viaskin® Peanut

SUMMARY:
This is an open label expanded access program for male and female patients 2 years or older, to provide continued desensitization treatment with DBV712 250 mcg.

DETAILED DESCRIPTION:
This study is an open-label Expanded Access Protocol to provide continued treatment with DBV712 for individuals completing a DBV clinical study. Participation is by invitation according to the inclusion criteria.

For individuals who have received DBV712 for longer than one year prior to entry into this protocol, where treatment allocation is unblinded, safety assessment and resupply of DBV712 will occur at 6-month intervals. There will be no other scheduled study visits. For individuals who have been on blinded treatment, a safety assessment will be conducted at Months 1 and 3. Visits for safety assessment and resupply of DBV712 will occur at 3-month intervals during the first 12 months. After a year, visits will occur at 6-month intervals. DBV712 will be supplied to participants at study visits to suffice until the next visit. For individuals who have been on blinded treatment, or off DBV712 treatment for more than 14 days prior to entry into this protocol, dosing consists of approximately 6 hours for the first week, 12 hours for the second week, then once daily, at approximately the same time of day.

Treatment with DBV712 will continue until, in the clinical judgement of the treating physician, the participant is no longer benefiting from continuation of the treatment, DBV712 is approved and available by prescription, or the study is terminated.

ELIGIBILITY:
Inclusion Criteria:

* Participation is by invitation, limited to individuals completing clinical study V712-303 (PEOPLE), previous Expanded Access Program or a DBV clinical study initiated after 31-Jan-2022
* Male and females; ages ≥ 2 years old at Visit 1 or current or prior studies.
* Negative urine pregnancy test for female participants of childbearing potential.

Exclusion Criteria:

* Early withdrawal from a DBV712 clinical study.
* History of non-compliance during the primary clinical study or unable to follow the protocol requirements.
* Generalized dermatologic disease extending widely on the skin.
* History of intolerance or who developed hypersensitivity to excipients of the DBV712 patches.

Ages: 2 Years to 17 Years | Sex: All
Age Groups: Child

CONTACTS AND LOCATIONS:
Locations (1):
- Early Access Care, LLC, Madison, Connecticut, United States